CLINICAL TRIAL: NCT00972595
Title: An Open-Label, Randomized, Single-Dose, 2-Period Crossover Study to Determine the Bioequivalence of 2 Formulations of Ondansetron in Healthy Young Adult Male and Female Subjects
Brief Title: Bioequivalence of Two Formulations of Ondansetron in Healthy Adults (0869-106)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0869-106; MK0869-106; 2009_657
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Ondansetron

ARMS (2):
- A (Experimental): clinical trial formulation
  Interventions: Drug: ondansetron clinical trial formulation
- B (Active Comparator): non-U.S. marketed formulation
  Interventions: Drug: ondansetron marketed formulation

INTERVENTIONS:
Drug: ondansetron clinical trial formulation — Single dose of an over-encapsulated 8 mg tablet of United Kingdom (U.K.) ondansetron (ZOFRAN™) in one of two treatment periods.
  Other Names: ZOFRAN™
  Arms: A
Drug: ondansetron marketed formulation — Single dose of an 8 mg tablet of U.K. ondansetron (ZOFRAN™) in one of two treatment periods.
  Other Names: ZOFRAN™
  Arms: B

SUMMARY:
This study will assess the bioequivalence of a Merck clinical trial formulation of ondansetron compared to a non-U.S. marketed formulation of ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* If female, subject is not pregnant or breast-feeding
* Subject has been a nonsmoker for at least 6 months
* Subject is in good health

Exclusion Criteria:

* Subject has a history of high blood pressure, asthma, other pulmonary disease, Gastrointestinal (GI) abnormalities/peptic ulcers, or cardiovascular, liver, neurologic, or kidney disease
* Subject is a habitual and heavy consumer of caffeine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2004-06; Primary Completion 2004-08 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- OE U.K. Tablet Then U.K. Tablet: Over-encapsulated (OE) United Kingdom (U.K.) tablet then U.K. tablet: Treatment OE U.K. tablet: an over-encapsulated single 8 mg tablet of United Kingdom (U.K.) ZOFRAN™ (ondansetron) taken orally/Treatment U.K. tablet: a single 8 mg tablet of ZOFRAN™ (ondansetron) which is marketed in the United Kingdom (U.K.) taken orally
- U.K. Tablet Then OE U.K. Tablet: U.K. tablet then OE U.K. tablet: Treatment U.K. tablet: a single 8 mg tablet of ZOFRAN™ (ondansetron) which is marketed in the United Kingdom (U.K.) taken orally/Treatment OE U.K. tablet: an over-encapsulated single 8 mg tablet of United Kingdom (U.K.) ZOFRAN™ (ondansetron) taken orally
Period: Period 1
Arm/Group | OE U.K. Tablet Then U.K. Tablet | U.K. Tablet Then OE U.K. Tablet
Started | 23 | 22
Completed | 22 | 22
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2
Arm/Group | OE U.K. Tablet Then U.K. Tablet | U.K. Tablet Then OE U.K. Tablet
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All Randomized Participants
Arm/Group | All Participants
Number analyzed (Participants) | 45
Age, Continuous [Mean (Full Range); unit: Years] | 34 [18 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 19
Height [Mean (Full Range); unit: Centimeters] | 170.8 [154.9 to 188.0]
Weight [Mean (Full Range); unit: Killograms] | 72.0 [45.5 to 102.7]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Area Under The Concentration Versus Time Curve (AUC(0-infinity)) For Ondansetron
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 24 hours postdose
Population: All 44 of the subjects who completed both Treatments OE U.K. tablet and U.K. tablet were included in the statistical analysis.
Measure: Least Squares Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- OE U.K. Tablet: Treatment OE U.K. tablet: an over-encapsulated single 8 mg tablet of United Kingdom (U.K.) ZOFRAN™ (ondansetron) taken orally
- U.K. Tablet: Treatment U.K. tablet: a single 8 mg tablet of ZOFRAN™ (ondansetron) which is marketed in the United Kingdom (U.K.) taken orally
Arm/Group | OE U.K. Tablet | U.K. Tablet
Number analyzed (Participants) | 44 | 44
ng*hr/mL | 257.8 (106.8) | 262.6 (105.6)
Statistical Analysis 1: Comparison: OE U.K. Tablet vs U.K. Tablet; Least-Squares Mean Ratio (OE U.K. tablet / U.K. tablet): an over-encapsulated single 8 mg tablet of United Kingdom (U.K.) ZOFRAN™ (ondansetron) taken orally; a single 8 mg tablet of ZOFRAN™ (ondansetron) which is marketed in the United Kingdom (U.K.) taken orally; Test type: Non-Inferiority or Equivalence — Study Primary Hypothesis: A single dose of the U.K. ZOFRAN™ (ondansetron) 8 mg tablet over-encapsulated is bioequivalent to a single dose of the U.K. ZOFRAN™ (ondansetron) 8-mg tablet. That is, the true geometric mean ratios (U.K. ZOFRAN™ tablet over-encapsulated/U.K. ZOFRAN™ tablet) of AUC0-∞ and Cmax for ondansetron each lie within the interval 0.80 to 1.25; Least-Squares Mean Ratio = 0.98, 90% CI [0.93 to 1.03]

2. Primary Outcome: Peak Plasma Concentration (Cmax) for Ondansetron
Time Frame: 24 hours post-dose
Population: All 44 of the subjects who completed both Treatment OE U.K. tablet and U.K. tablet were included in the statistical analysis.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | OE U.K. Tablet | U.K. Tablet
Number analyzed (Participants) | 44 | 44
ng/mL | 41.3 (13.7) | 41.8 (13.6)
Statistical Analysis 1: Comparison: OE U.K. Tablet vs U.K. Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Study Primary Hypothesis: A single dose of the U.K. ZOFRAN™ (ondansetron) 8 mg tablet over-encapsulated is bioequivalent to a single dose of the U.K. ZOFRAN™ (ondansetron) 8 mg tablet. That is, the true geometric mean ratios (U.K. ZOFRAN™ tablet over-encapsulated/U.K. ZOFRAN™ tablet) of AUC0-∞ and Cmax for ondansetron each lie within the interval 0.80 to 1.25; Least-Squares Mean Ratio = 0.99, 90% CI [0.93 to 1.05]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were captured from Treatment Period 1, Day 1 to 14 days Post Last Dose of Study Drug in Treatment Period 2, including the 7 day washout in between periods
Arm/Group | OE U.K. Tablet Then U.K. Tablet | U.K. Tablet Then OE U.K. Tablet
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/22
Other Adverse Events (participants affected / at risk) | 13/45 | 6/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OE U.K. Tablet Then U.K. Tablet (N=23) | U.K. Tablet Then OE U.K. Tablet (N=22)
Aborted Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OE U.K. Tablet Then U.K. Tablet (N=45) | U.K. Tablet Then OE U.K. Tablet (N=44)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Ear Infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Haematocrit Decreased (Investigations) | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 7 | 5
Sinus Headache (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.